CLINICAL TRIAL: NCT07186023
Title: Intervention Evaluation for Late-life Depression in Taiwan Urban and Rural Areas: Long-term Tracking and Prediction of Non-pharmaceutical Interventions by Smart AI Technologies
Brief Title: Effects of Mindfulness or Brain Stimulation Intervention for Late-life Adults in Taiwan Urban and Rural Areas
Acronym: PredictNPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Ai-Ling Hsu, Assistant Investigator, National Health Research Institutes, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: EC1140405; CG-114-GP-23 (Other Grant/Funding Number: National Health Research Institutes)
Record Dates: First submitted 2025-08-14; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Late-Life Adults; Late-Life Prodromal Depression; Late-Life Depression; Mindfulness; Brain Stimulation Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- MBSR (Active Comparator): Mindfulness-Based Stress Reduction
  Interventions: Behavioral: MBSR
- MBWC (Active Comparator): Mindfulness-Based Well-Being Curriculum
  Interventions: Behavioral: MBWC
- MBCI (Active Comparator): Mindfulness-Based Curriculum for Insomnia
  Interventions: Behavioral: MBCI
- BSI (Other): Brain Stimulation Intervention
  Interventions: Device: BSI

INTERVENTIONS:
Behavioral: MBSR — Mindfulness-Based Stress Reduction
  Arms: MBSR
Behavioral: MBWC — Mindfulness-Based Well-Being Curriculum
  Arms: MBWC
Behavioral: MBCI — Mindfulness-Based Curriculum for Insomnia
  Arms: MBCI
Device: BSI — Brain Stimulation Intervention
  Arms: BSI

SUMMARY:
This randomized controlled trial will examine the effects of mindfulness-based interventions and brain stimulation interventions on cognitive function and psychological well-being in older adults. The study will employ a comprehensive assessment approach incorporating psychological evaluations, behavioral assessments, psychophysiological measurements, and neuroimaging analyses to characterize the outcome of nonpharmaceutical interventions in improving geriatric well-being or reducing depression severity.

ELIGIBILITY:
Inclusion Criteria for individuals participating in mindfulness-based Interventions:

* Literate or have received an education above the elementary level.
* Have normal or corrected vision and hearing, able to communicate and understand explanations.
* Right-handed individuals as assessed by the Edinburgh Handedness Inventory.

Exclusion Criteria for individuals participating in mindfulness-based Interventions:

* Individuals with dementia, stroke, cerebrovascular disease, brain injury, epilepsy, or Parkinson's disease.
* Individuals with neurological system disorders.
* Individuals with alcohol or drug dependence.
* Individuals with other major physical illnesses, such as diabetes, heart failure, or endocrine abnormalities, or those who have experienced an acute myocardial infarction within the past three months.
* Individuals with metal objects in the body that cannot undergo magnetic resonance imaging (MRI), such as cardiac pacemakers, vascular clips, hearing aids, artificial joints, steel pins, etc.
* Individuals with Claustrophobia.
* Individuals in pregnancy or possibility of pregnancy.

Inclusion Criteria for individuals participating in brain stimulation Intervention:

* Individuals diagnosed with major depressive disorder by psychiatrists according to the Diagnostic and Statistical Manual, and who can cooperate with the psychiatric outpatient clinic regulations.
* Literate or have received an education above the elementary level.
* Have normal or corrected vision and hearing, able to communicate and understand explanations.
* Right-handed individuals as assessed by the Edinburgh Handedness Inventory.
* Individuals are prescribed brain stimulation therapy by clinical physicians.

Exclusion Criteria for individuals participating in brain stimulation Intervention:

* Individuals with dementia, stroke, cerebrovascular disease, brain injury, epilepsy, or Parkinson's disease.
* Individuals with neurological system disorders.
* Individuals with alcohol or drug dependence.
* Individuals with other major physical illnesses, such as diabetes, heart failure, or endocrine abnormalities, or those who have experienced an acute myocardial infarction within the past three months.
* Individuals with metal objects in the body that cannot undergo magnetic resonance imaging (MRI), such as cardiac pacemakers, vascular clips, hearing aids, artificial joints, steel pins, etc.
* Individuals with Claustrophobia.
* Individuals in pregnancy or possibility of pregnancy.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes in neural activation related to emotional processing, sensory processing, attention, and memory-related brain regions. | Baseline assessment conducted during the 4-week period prior to intervention initiation; follow-up assessment conducted during the 4-week period following intervention completion.
  Significant alterations in blood oxygen level-dependent (BOLD) signal amplitude during task-based functional magnetic resonance imaging (fMRI).
Changes in resting-state functional connectivity within and between brain networks | Baseline assessment conducted during the 4-week period prior to intervention initiation; follow-up assessment conducted during the 4-week period following intervention completion.
  Statistically significant alterations in intrinsic functional connectivity parameters derived from blood-oxygen-level-dependent (BOLD) signals acquired during resting-state functional magnetic resonance imaging (rs-fMRI).

SECONDARY OUTCOMES:
Regional brain morphometric changes, assessed by quantitative analysis of gray matter volume, thickness, and density differences using high-resolution structural magnetic resonance imaging. | Baseline assessment conducted during the 4-week period prior to intervention initiation; follow-up assessment conducted during the 4-week period following intervention completion.
  Statistically significant alterations in regional gray matter volume (measured in cubic millimeters), thickness (measured in millimeters) or density (represented as a percentage between 0 and 1) compared to baseline measurements.
Self-reported neuropsychological outcomes assessed through validated Wechsler Adult Intelligence Scale (WAIS). | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Statistically significant changes across 3 time points using WAIS across subsets of facial memory test and (scores between 0 and 48), digit span in forward (scores between 0 and 16) and backward order (scores between 0 and 14), block design (scores between 0 and 68), digit symbol-coding (scores between 0 and 133).
Scores of the total number of category-naming items correctly named within one minute for testing verbal fluency. | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Statistically significant changes across 3 time points using Verbal fluency scores in categories of colors, animals, cities, and fruits.
Changes in the depression scale | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Depression scale changes measured by the geriatric depression scale (scores between 0 and 15) and the 17-item Hamilton depression rating scale (scores between 0 and 52) across 3 time points.
Changes in anxiety scale | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Anxiety scale changes measured by the Hamilton anxiety rating scale (scores between 0 and 48) across 3 time points.
Changes in the loneliness scale | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Changes of the loneliness scale developed by the University of California, Los Angeles, across 3 time points
Changes in perceived stress | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Changes of the 14-item perceived stress scale (scores between 0 and 56) across 3 time points
Changes in the apathy scale | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Changes of the 18-item apathy evaluation scale (scores between 0 and 72) across 3 time points
Changes in self-reported sleep outcomes assessed through sleepiness and sleep quality | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Changes of the 3-item insomnia severity index for sleepiness (scores between 0 and 28) and the 10-item Pittsburgh Sleep Quality Index for sleep quality across 3 time points
Changes in self-reported intervention outcomes in terms of mindfulness, flourishing, and well-being | Baseline (within 4 weeks pre-intervention), immediate post-intervention (within 1 week of completion), and 1-month follow-up (within 1 week of the 1-month milestone).
  Changes of Intervention outcomes assessed by the 39-item five-facet mindfulness questionnaire, 30-item flourishing scale across 5 domains (mercifulness, playfulness, respectfulness, peacefulness, healthfulness), and two forms of well-being scale (short and long forms) across 3 time points. The short form is the World Health Organization-five well-being index (scores between 0 and 25). The long form is a 29-item well-being scale for the elderly in Taiwan (scores between 0 and 145).
Dynamic patterns of objective sleep parameters assessed through smart watch monitoring | Continuous physiological monitoring conducted from 4 weeks pre-intervention through 4 weeks post-completion of the 1-month follow-up period (total monitoring duration: 16 weeks).
  Dynamic patterns of sleep indices (including sleep stage duration, sleep onset latency, and sleep efficiency), measured by a smart watch from baseline through to 1-month follow-up assessments.
Dynamic patterns of objective cardiovascular parameters assessed through smart watch monitoring | Continuous physiological monitoring conducted from 4 weeks pre-intervention through 4 weeks post-completion of the 1-month follow-up period (total monitoring duration: 16 weeks).
  Dynamic patterns of indices deriving from heart rate (including heart rate variability and stress), measured by a smart watch, from baseline through to 1-month follow-up assessments.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Shuang Ho Biomedical Park, Taipei Medical University, New Taipei City
  - National Center for Geriatrics and Welfare Research, Yunlin

IPD SHARING:
Plan to Share IPD: No